CLINICAL TRIAL: NCT04874857
Title: The Effect of Aromatherapy Massage Applied to Hemodialysis Patients With Muscle Cramp on Cramp Frequency, Severity of Pain and Quality of Life
Brief Title: The Effect of Aromatherapy Massage Applied to Hemodialysis Patients With Muscle Cramp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Serife Cetin, PhD student, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Erciyes University; PhD student (Other: Erciyes University)
Record Dates: First submitted 2021-04-21; First posted 2021-05-06 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Muscle Cramps; Aromatherapy; Hemodialysis; Quality of Life; Pain
MeSH Terms: conditions — Muscle Cramp; Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group (Aromatherapy group) (Experimental): With a mixture of Lavandula angustifolia, Rosmarinus officinalis L. and Origanum majorana L. essential oils, the foot and lower leg will be massaged for three sessions a week for 30 minutes in each session for four weeks.
  Interventions: Other: Lavandula angustifolia, Rosmarinus officinalis L. and Origanum majorana L.
- Placebo group (Experimental): The foot and lower leg will be massaged with baby oil for four weeks, three sessions a week, 30 minutes in each session.
  Interventions: Other: Baby oil
- Control group (No Intervention): No application will be made in addition to standard HD treatment.

INTERVENTIONS:
Other: Lavandula angustifolia, Rosmarinus officinalis L. and Origanum majorana L. — Massage application
  Arms: Intervention group (Aromatherapy group)
Other: Baby oil — Massage application
  Arms: Placebo group

SUMMARY:
This study is a randomized controlled and single-blind study consisting of qualitative and quantitative stages to evaluate the effect of aromatherapy massage on cramp frequency, cramp pain severity and quality of life in crampy hemodialysis (HD) patients.

DETAILED DESCRIPTION:
Data-collecting interviewers are blind to which patients are in which group. The days and sessions of the groups were randomly determined after patients meeting the research criteria of the intervention, placebo control, and control groups were ranked.

The population of the study consists of 566 patients treated in institutions that allow the research to be conducted.

145 patients participated in the study and the study was terminated with 94 patients. In the study, aromatherapy massage was applied to the intervention group, baby oil massage was applied to the placebo control group, while no application was made to the control group other than routine care. Aromatherapy massage to the intervention group; It was applied with a mixture of 7% lavender, rosemary and marjoram essential oils.

Dependent Variables: Cramp frequency, mean cramp pain severity, and quality of life scale total score.

Independent Variables: age, gender, body mass index, marital status, educational status, income level, sociodemographic characteristics such as smoking and alcohol use, characteristics related to the diagnosis-treatment process, concomitant diseases and laboratory parameters.

Research data; Intervention and Placebo Group Situation Evaluation Chart, Personal Information Form, Personal Interview Form, Visual Analogue Scale, Quality of Life Index Dialysis Version-III and Control, Intervention and Placebo Group Monitoring Chart were collected. The qualitative data obtained in the study were evaluated using descriptive and content analysis methods. Statistical Package for the Social Sciences program was used to evaluate the quantitative data. A value of p < 0.05 will be accepted as statistical significance criterion. In order to carry out the study, the necessary Academic Committee decision, Ethics Committee approval (dated 11 November 2020 and numbered 13) and institutional permission were obtained. The individuals included in the study were informed about the purpose of the study.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old,
* Able to answer questions and communicate,
* Is conscious and does not have a mental problem,
* Speaks Turkish,
* No hearing, sight or speech impairment,
* Having HD treatment for at least six months,
* Receiving three HD treatment sessions a week,
* Dialysis with bicarbonate dialysate,
* Kt / V value> 1.2,
* Having a constant dry weight for the last month,
* Experiencing cramps during hemodialysis sessions or at any other time and who scored at least three or more when the severity of cramp pain was evaluated with the Visual Analog Scale (VAS),
* Patients who are not allergic to the oils used for massage will be included in the study.

Exclusion Criteria:

* Pregnant and breastfeeding women,
* Cancer,
* Diabetic foot,
* Lower extremity amputation,
* Having neurological diseases such as epilepsy, parkinson, dementia, Alzheimer,
* Those with paraplegia,
* The lower leg is in a size that prevents the application of massage,
* had surgery in the last three months,
* Loss of sensation more than 50% due to neuropathy due to various reasons,
* Open wound in the foot and lower leg, infection, necrosis, fracture / fracture suspected, soft tissue damage, burn,
* Peripheral vascular disease,
* Deep vein thrombosis,
* Receiving treatment to prevent cramping,
* Having a severe electrolyte (such as potassium, magnesium, calcium) disorder in blood values,
* Patients using any of the complementary and integrated methods in the last month will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scala (VAS) | During 1 month
  The widespread use of VAS, which has been used in the research of subjective concepts from past years to the present, has been realized after in 1969. This scale; There is a number value of "0 (no pain)" at the beginning and "10 (the most unbearable pain)" at the end. The patient marks the severity of the cramp he is experiencing at that moment, and the starting and ending points of the scale as criteria. A VAS value between 1-3 means "mild pain", between 4-6 means "moderate pain", and a value between 7-10 means "severe pain". Participants will mark the scale each time they experience a cramp.

SECONDARY OUTCOMES:
Quality of Life Index Dialysis Version - III | At the first and last meeting in 1 month
  "Quality of Life Index Dialysis Version-3" was developed in 1985 in America. This scale consists of two parts measuring satisfaction from different areas of life and the importance of these areas for the individual, each part contains 34 items. In the satisfaction part of the 6-degree Likert-type scale consisting of 64 items, there are expressions from "very satisfied" to "not satisfied at all", and "very important to very unimportant" in the importance part. The scale has 4 sub-dimensions: health and function, socio-economic, psychological-beliefs, and family. The "translated total score" is obtained by combining the satisfaction and importance scores of the scale with a special formula.

CONTACTS AND LOCATIONS:
Overall Officials: Serife Cetin, PhD, Principal Investigator — Kayseri University
Locations (1):
- Erciyes University, Melikgazi, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No